CLINICAL TRIAL: NCT00123851
Title: A Phase II Study of OSI-774 (Tarceva) in Combination With Oxaliplatin and Capecitabine in Previously Treated Patients With Stage IV Colorectal Cancer
Brief Title: Tarceva, Capecitabine and Oxaliplatin for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Sanofi-Synthelabo (Industry); OSI Pharmaceuticals (Industry); Hoffmann-La Roche (Industry); Genentech, Inc. (Industry); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-269
Record Dates: First submitted 2005-07-25; First posted 2005-07-26 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis
Keywords: Colorectal; Metastatic Colorectal Cancer; Oxaliplatin; Tarceva; Capecitabine; Xeloda
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Erlotinib Hydrochloride; Capecitabine; Oxaliplatin

INTERVENTIONS:
Drug: Tarceva (OSI-774)
Drug: Capecitabine
Drug: Oxaliplatin

SUMMARY:
This trial is designed to investigate the safety, tolerability and the effectiveness when OSI-774 (tarceva) is combined with oxaliplatin and capecitabine in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Patients will be treated with OSI-774 (orally) daily, oxaliplatin (intravenously) every 3 weeks, and capecitabine (orally) twice daily for 14 days followed by a 7-day rest period. This will constitute a 21-day treatment cycle. Treatment will continue until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Patients with histologic proof of adenocarcinoma of the colon or rectum (colorectal carcinoma) with evidence of metastatic disease.
* Patients must have received one (and only 1) prior chemotherapy regimen for metastatic disease. Patients who received adjuvant therapy and then 1 regimen for metastatic disease are eligible. Patients who received adjuvant therapy and recur within 12 months of completion of adjuvant therapy are also eligible.
* Patients who have received prior radiation therapy, either in the adjuvant or metastatic setting, for colorectal carcinoma.
* All of the following must apply:

  * Greater than 4 weeks must have elapsed from the time of major surgery and patients must have recovered from the effects (e.g., laparotomy); *Greater than 2 weeks must have elapsed from the time of minor surgery and patients must have recovered from the operation. (Insertion of a vascular access device is not considered major or minor surgery.);
  * Greater than 4 weeks must have elapsed from the time of major radiotherapy [RT] (e.g., chest or bone palliative RT);
  * Greater than 4 weeks must have elapsed from the completion of previous chemotherapy and patients must have recovered from any related toxicities;
  * Greater than 4 weeks must have elapsed from the participation in any investigational drug study.
* ECOG performance status < 2 ; life expectancy > 12 weeks
* Patients must have normal organ and marrow function as defined below:

ANC > 1500/mm3; hemoglobin > 9.0 gm/dl; platelets > 100,000/mm3; SGOT < 2.5x upper limits of normal if no evidence of liver metastases or < 5x upper limits of normal if evidence of liver metastases; total bilirubin < 1.5x upper limits of normal; Alk Phos < 2.5x upper limits of normal (or < 5x upper limits of normal if evidence of liver metastases or < 10x upper limits of normal if evidence of bone disease).

Exclusion Criteria:

* Patients with peripheral neuropathy of grade 2 or greater severity.
* Uncontrolled high blood pressure.
* Unstable angina.
* Symptomatic congestive heart failure.
* Myocardial infarction < 12 months prior to registration.
* Serious uncontrolled cardiac arrhythmia.
* New York Heart Association classification III or IV.
* Active or uncontrolled infection.
* Medical or psychiatric conditions which, in the opinion of the investigator, make participation in an investigational trial of this nature a poor risk.
* Patients with known brain metastases or carcinomatous meningitis should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* No concurrent malignancy of any site, except for limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration and agree to use an effective method of contraception.
* Patients who are pregnant or lactating.
* Patients with prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil.
* Patients previously treated with oxaliplatin, OSI-774 or another epidermal growth factor inhibitor (EGFR).
* Patients lacking physical integrity of the upper gastrointestinal tract.
* Patients with other serious uncontrolled medical conditions that the investigator feels might compromise study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2003-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine the response rate of OSI-774 when given in combination with oxaliplatin and capecitabine in patients with previously-treated locally advanced, locally recurrent, or metastatic colorectal adenocarcinoma

SECONDARY OUTCOMES:
To assess overall survival, progression-free survival, time to progression and duration of response
To evaluate the toxicities of the combination of OSI-774, oxaliplatin and capecitabine in this population of patients with colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Meyerhardt, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Meyerhardt JA, Zhu AX, Enzinger PC, Ryan DP, Clark JW, Kulke MH, Earle CC, Vincitore M, Michelini A, Sheehan S, Fuchs CS. Phase II study of capecitabine, oxaliplatin, and erlotinib in previously treated patients with metastastic colorectal cancer. J Clin Oncol. 2006 Apr 20;24(12):1892-7. doi: 10.1200/JCO.2005.05.3728. PMID 16622264